CLINICAL TRIAL: NCT04768075
Title: Randomized, Double-blind, Placebo-controlled, Multi-center Study of Camrelizumab Combined With SRT/WBRT and Chemotherapy in Patients of NSCLC With Brain Metastases of Driven Gene-negative and Not Received Systemic Chemotherapy
Brief Title: Camrelizumab Combined With SRT/WBRT and Chemotherapy in Patients With Brain Metastases of Driven Gene-negative NSCLC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangdong Association of Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTONG2003
Record Dates: First submitted 2021-02-04; First posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Non-Small-Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — camrelizumab; Cisplatin; Carboplatin; Pemetrexed; Paclitaxel; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Camrelizumab group (Experimental): subject will receive Camrelizumab intravenously(IV) PLUS pemetrexed or paclitaxel or albumin paclitaxel PLUS cisplatin or carboplatin AUC 5 on Day 1 of each 3-week cycle(Q3W) for 4-6 cycles followed by Camrelizumab ± pemetrexed IV Q3W until progression (up to approximately 2 years).
  Whether the subject accepts intracranial radiotherapy will be decided by investigators according to the guidelines and the conditions of the subjects.
  Interventions: Drug: Camrelizumab; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed; Drug: Paclitaxel; Drug: Albumin paclitaxel
- placebo group (Placebo Comparator): subject will receive placebo intravenously (IV) PLUS pemetrexed or paclitaxel or albumin paclitaxel PLUS cisplatin or carboplatin AUC 5 on Day 1 of each 3-week cycle(Q3W) for 4-6 cycles followed by placebo ± pemetrexed IV Q3W until progression (up to approximately 2 years).
  Whether the subject accepts intracranial radiotherapy will be decided by investigators according to the guidelines and the conditions of the subjects.
  Interventions: Drug: Placebo; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed; Drug: Paclitaxel; Drug: Albumin paclitaxel

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab is a humanized anti-PD1 IgG4 monoclonal antibody
  Other Names: SHR-1210
  Arms: Camrelizumab group
Drug: Placebo — IV infusion Simulator of Camrelizumab
  Other Names: Simulator of Camrelizumab
  Arms: placebo group
Drug: Cisplatin — IV infusion
  Other Names: cisplatinum
Drug: Carboplatin — IV infusion
  Other Names: Carboplat
Drug: Pemetrexed — IV infusion
  Other Names: Pemetrexed disodium
Drug: Paclitaxel — IV infusion
  Other Names: Paclitaxel injection
Drug: Albumin paclitaxel — IV infusion
  Other Names: Nab-paclitaxel

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, multi-center clinical study. Target population is patients with stage IV non-small cell lung cancer who had not received systemic chemotherapy. Study objective is to compare the efficacy and safety of Camrelizumab + carboplatin/cisplatin + pemetrexed /paclitaxel / albumin paclitaxel ± SRT/WBRT with placebo + carboplatin/cisplatin + pemetrexed /paclitaxel / albumin paclitaxel ± SRT/WBRT. Camrelizumab is a humanized anti-PD1 IgG4 monoclonal antibody.

DETAILED DESCRIPTION:
Detailed Description:

In this study, eligible subject will be randomized into study arm or control arm to accept study treatment. Paticipant was confirmed without EGFR activating mutation or ALK fusion and received no prior systemic therapy. Patients would receive Camrelizumab/placebo in combination with chemotherapy for 4-6 cycles，non-squamous subject followed by Camrelizumab/placebo + pemetrexed as maintenance treatment until progression or unacceptable toxicity, squamous subject followed by Camrelizumab/placebo as maintenance treatment until progression or unacceptable toxicity, Camrelizumab/placebo for a maximum of 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological diagnosis of non-small cell lung cancer（NSCLC）;
2. MRI confirmed brain parenchyma metastasis, ≥ 3 brain lesions, or 1-2 brain lesions but not suitable for local treatment or refused local treatment. At least one brain measurable lesion ≥ 5mm . Included with or without neurological symptoms;
3. Has not received prior systemic treatment for metastatic NSCLC. Subjects who have received prior neo-adjuvant, adjuvant chemotherapy, or chemoradiotherapy with curative intent must have experienced interval of at least 12 months from diagnosed of advanced or metastatic disease since the end of surgery;
4. Has confirmation that epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK)-directed therapy is not indicated;
5. Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status;
6. Has adequate organ function;
7. Women of childbearing age must undergo a serological pregnancy test within 7 days before the first dose with negative results. Subjects willing to use an effective contraceptive method during the study and within 90 days after the last dose of study medication;
8. Subjects should be able to follow the research and follow-up procedures;
9. Subjects should be voluntarily participating in clinical studies and informed consent should be signed;

Exclusion Criteria:

1. Brain metastases with hemorrhage；
2. Meningeal involvement with metastatic carcinoma;
3. Subjects with ROS1 mutation, RET fusion positive, BRAF V600E mutation, NTRK fusion positive;
4. Participated in other clinical trials, or finish other clinical trials within 4 weeks;
5. Subject was received irradiation of brain;
6. Subjects have received solid organ or blood system transplantation;
7. Active autoimmune diseases requiring systemic treatment (such as the use of disease remission drugs, corticosteroids or immunosuppressants) occurred within 2 years before the first administration. Alternative therapy (such as thyroxine, insulin or physiological corticosteroids for adrenal or pituitary insufficiency) is not considered systemic therapy;
8. Subjects diagnosed immunodeficiency or receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy of non-related tumor within 7 days before the first dose; allowed physiological dose of glucocorticoid (≤10 mg/day Prednisone or equivalent);
9. Within 1 year before the first dose, there was a history of non-infectious pneumonia or interstitial lung disease requiring glucocorticoid treatment;
10. Subjects with grade II or above myocardial ischemia or myocardial infarction and poorly controlled arrhythmias (QTc interval > 450 ms for males and QTc interval > 470 ms for females). Subjects with grade III-IV cardiac insufficiency or with left ventricular ejection fraction (LVEF) less than 50% according to NYHA criteria;
11. Has known history of Human Immunodeficiency Virus (HIV)；
12. Untreated active hepatitis B；
13. Subjects have active hepatitis B；
14. Subjects have severe infections within 4 weeks of the first dose of study treatment；
15. Subjects with clinically significant bleeding symptoms or with obvious bleeding tendency in the first month;
16. Women who are pregnant or lactating；
17. Has known allergy to Camrelizumab, or pemetrexed, or paclitaxel, or albumin paclitaxel, or carboplatin, or cisplatin or any of accessories;
18. A prior malignancy other than NSCLC within 5 years before randomization，except carcinoma in situ of the cervix or basal cell carcinoma or squamous cell carcinoma of skin cancer with adequately treated, localized prostate cancer or ductal carcinoma in situ after radical resection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-03-05 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Intracranial Progression-Free Survival(iPFS) | up to 24 month
  Intracranial Progression-free survival is defined as the duration from date of enrollment to the first occurrence of progression in brain metastasis disease or death from any cause or switch therapy

SECONDARY OUTCOMES:
Intracranial Objective Response Rate (iORR) | up to 24 month
  iORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response(PR: ≥30% decrease in the sum of diameters of target lesions) in brain lesion per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Objective Response Rate (ORR) | up to 24 month
  ORR was defined as the percentage of participants in the analysis population who had a CR or a PR.
Progression-Free Survival (PFS) | up to 24 month
  PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first.
Overall Survival (OS) | up to 24 month
  OS was defined as the time from randomization to death due to any cause.
Duration of Response (DOR) | up to 24 month
  DOR was defined as the time from first documented evidence of a CR or PR until PD or death
Quality of Life (QoL) | up to 24 month
  Evaluate according to the quality of life score V3.0，higher scores mean a better outcome.
Adverse events (AEs)/ Serious adverse event (SAE) | up to 24 month
  All adverse event/Serious adverse event that occurred during the study period according to CTCAE v 5.0
Simple Mental State Scale of Intelligence (MMSE) | up to 24 month
  Assessment of cognitive function based on the MMSE ,the values from 0 to 30, higher scores mean a better outcome.
Revised Hopkins Vocabulary Learning Test Scale (HVLT-R) | up to 24 month
  Assessment of cognitive function based on the HVLT-R，higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Wu Yi Long, PhD, Principal Investigator — Guangdong Lung Cancer Institute, Guangdong General Hospital, Guangdong Academy of Medical Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li YS, Yu Q, Bu Q, Lin L, Ning F, Zhao Y, Wu G, Lin G, Zang A, Sun H, Huang J, Tu HY, Ma S, Zhou C, Liu A, Wang C, Yao Y, Han G, Zhao J, Zhou Q, Yan HH, Liu SM, Zheng MM, Lv J, Cheng F, Chen Z, Zhong WZ, Pan Y, Yang JJ, Wu YL. First-Line Camrelizumab Versus Placebo Plus Chemotherapy With or Without Radiotherapy for Brain Metastases in NSCLC: The CTONG 2003 Randomized Placebo-Controlled Trial. J Thorac Oncol. 2025 Jul;20(7):928-940. doi: 10.1016/j.jtho.2025.02.004. Epub 2025 Feb 8. PMID 39929333